CLINICAL TRIAL: NCT01560507
Title: Tailored Smoking Cessation Treatment for LIVE FOR LIFE® Participants
Acronym: LiveForLife2
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Low Recruitment
Sponsor: Duke University (Other)
Collaborators: Philip Morris USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00032605
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Results first posted 2013-11-19 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-11

CONDITIONS: Cigarette Smoking; Nicotine Dependence
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Disorder | interventions — Varenicline; Bupropion; Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- varenicline (Chantix) (Active Comparator): This group will consist of smokers who, based on smoking behavior, DO NOT respond favorably to pre-cessation Nicotine Replacement Therapy (NRT) assessed the day before the scheduled quit day. They will receive varenicline.
  Interventions: Drug: varenicline (Chantix)
- nicotine patches (Active Comparator): This group will consist of smokers who, based on smoking behavior, respond favorably to pre-cessation NRT (assessed the day before the scheduled quit day). They will continue to using only nicotine patches.
  Interventions: Drug: nicotine patches
- bupropion (Zyban) and nicotine patches (Active Comparator): This group will consist of smokers who, based on smoking behavior, DO NOT respond favorably to pre-cessation NRT (assessed the day before the scheduled quit day). They will receive bupropion with nicotine patches.
  Interventions: Drug: bupropion (Zyban); Drug: nicotine patches

INTERVENTIONS:
Drug: varenicline (Chantix) — For the first 3 days after being switched from NRT (occurring at one week before the rescheduled quit date), smokers in this group will receive varenicline at a dose of 0.5 mg once per day followed by 0.5 mg twice a day for the remaining 4 days of that week. Subsequently, the dose will be 1 mg twice per day, and will remain at that dose for the remainder of the 12 weeks.
  Other Names: Chantix; varenicline
  Arms: varenicline (Chantix)
Drug: bupropion (Zyban) — After being switched from NRT (occurring at one week before the rescheduled quit date), smokers in this group will receive 150mg of bupropion once daily and 21mg nicotine patch for first 3 days; 150mg of bupropion twice daily and 21mg nicotine patch for 7 weeks; 150mg of bupropion twice daily and 14mg nicotine patch for 2 weeks and 150mg of bupropion twice daily and 7mg nicotine patch for 2 weeks.
  Other Names: Zyban; bupropion
  Arms: bupropion (Zyban) and nicotine patches
Drug: nicotine patches — 21mg nicotine patch for first 11 weeks; 14mg nicotine patch for next 2 weeks; 7mg nicotine patch for final 2 weeks.
  Arms: bupropion (Zyban) and nicotine patches; nicotine patches

SUMMARY:
The purpose of this study is to ascertain: 1) the rate of smoking cessation obtained using an adaptive treatment algorithm developed in previous clinical trials, in order to calculate cost-effectiveness of the treatment; 2) the relationship between genotype and response to cigarette smoking cessation treatment.

DETAILED DESCRIPTION:
Previous research has shown that the initial response to nicotine patch treatment can be used to decide whether the patch alone is likely to help smokers to quit or whether alternative prescription medications may be needed to achieve smoking abstinence. This study applies the knowledge gained from this previous research to adapt the smoking cessation treatment provided to participants, based on their degree of smoking reduction during the first four weeks of nicotine patch treatment. By demonstrating effectiveness of this algorithm, this study may lead to further dissemination of the adaptive treatment strategy to other health care settings. Additionally, by gathering further information relating genomic markers to outcome, the foundation will be laid for potential practical application of this index in other settings.

ELIGIBILITY:
Inclusion Criteria:

* Duke employees who are enrolled in a Duke Health Plan and intend to remain employed at Duke for the next six months;
* Dependents of Duke employees who meet the above criteria;
* 18-65 years old;
* Currently smoke an average of at least 10 cigarettes per day;
* Willing to take Chantix or Zyban;
* Express a desire to quit smoking within the next 30 days.

Exclusion Criteria:

* Hypertension;
* Hypotension with symptoms (systolic <90 mm Hg, diastolic <60 mm Hg);
* Coronary heart disease;
* Lifetime history of heart attack;
* Cardiac rhythm disorder (irregular heart rhythm);
* Chest pains (unless history, exam, and ECG clearly indicate a non-cardiac source);
* Cardiac (heart) disorder (including but not limited to valvular heart disease, heart murmur, heart failure);
* Extensive active skin disorder;
* Liver or kidney disorder (except kidney stones, gallstones);
* Gastrointestinal disease other than gastroesophageal reflux or heartburn;
* Active ulcers in the past 30 days;
* Currently symptomatic lung disorder/disease (including but not limited to COPD, emphysema, and asthma);
* Brain abnormality (including but not limited to stroke, brain tumor, and seizure disorder);
* Migraine headaches that occur more frequently than once per week;
* Recent, unexplained fainting spells;
* Diabetes treated with insulin; non-insulin treated diabetes (unless glucose is less than 180mg/dcl and HbA1c is less than 7%);
* Current cancer or treatment for cancer in the past six months (except basal or squamous cell skin cancer);
* Other major medical condition;
* Suicidal ideation (within the past 10 years) or lifetime occurrence of attempted suicide;
* Pregnant or nursing mothers;
* Current psychiatric disease (with the exception of anxiety disorders, OCD and ADHD);
* Current depression;
* Bulimia or anorexia;
* Alcohol abuse;
* Significant adverse reaction to bupropion/Wellbutrin/Zyban, Chantix/Varenicline or nicotine patches in the past.
* Use (within the past 30 days) of:

  * Wellbutrin, bupropion, Zyban, Chantix, nicotine replacement therapy or any other smoking cessation aid.
  * Medications that are known to affect smoking cessation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed E Rose, Ph.D., Principal Investigator — Duke University
Locations (2):
- United States (2):
  - Duke Center forSmoking Cessation, Durham, North Carolina
  - Duke Center for Smoking Cessation, Raleigh, North Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from May 2012 until May 2013. We were only able to enter 19 of the 300 subjects into the study. We discontinued the study in July 2013 because of the recruitment difficulties.
Pre-assignment Details: Of the 19 subjects who signed a consent form: 9 subjects began study participation; 7 subjects were excluded prior to receiving study drug because of medical issues and 3 subjects met other exclusion criteria and were excluded prior to receiving study drug.
Groups:
- Varenicline (Chantix): This group consists of smokers who, based on smoking behavior, DO NOT respond favorably to pre-cessation NRT (assessed the day before the scheduled quit day). They received varenicline.
- Nicotine Patches: This group consists of smokers who, based on smoking behavior, respond favorably to pre-cessation NRT (assessed the day before the scheduled quit day). They continued to use only nicotine patches.
- Bupropion (Zyban) and Nicotine Patches: This group consists of smokers who, based on smoking behavior, DO NOT respond favorably to pre-cessation NRT (assessed the day before the scheduled quit day). They received bupropion and nicotine patches.
Period: Overall Study
Arm/Group | Varenicline (Chantix) | Nicotine Patches | Bupropion (Zyban) and Nicotine Patches
Started | 5 | 2 | 2
Completed | 1 | 0 | 0
Not Completed | 4 | 2 | 2
Not completed — Lost to Follow-up | 3 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline (Chantix) | Nicotine Patches | Bupropion (Zyban) and Nicotine Patches | Total
Number analyzed (Participants) | 5 | 2 | 2 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 2 | 9
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.02 (10.75) | 33.47 (0.43) | 39.61 (3.94) | 42.36 (9.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 5
  Male | 2 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 5 | 2 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: Cost-effectiveness of the Adaptive Treatment Approach to Smoking Cessation
Description: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Time Frame: End of study drug treatment period (11-12 weeks)
Arm/Group | Varenicline (Chantix) | Nicotine Patches | Bupropion (Zyban) and Nicotine Patches
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Quit Success Genotype Score
Description: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed."
Time Frame: After 6 month Follow-Up
Population: Study was terminated early due to difficulties with enrollment. No outcome measures were assessed.
Groups:
- Bupropion (Zyban) and Nicotine Patches: This group consists of smokers who, based on smoking behavior, DO NOT respond favorably to pre-cessation NRT (assessed the day before the scheduled quit day). They received bupropion and nicotine patches.
  bupropion (Zyban) & nicotine patches: After being switched from NRT (occurring at one week before the rescheduled quit date), smokers in this group will receive 150mg of bupropion once daily and 21mg nicotine patch for first 3 days; 150mg of bupropion twice daily and 21mg nicotine patch for 7 weeks; 150mg of bupropion twice daily and 14mg nicotine patch for 2 weeks and 150mg of bupropion twice daily and 7mg nicotine patch for 2 weeks.
Arm/Group | Varenicline (Chantix) | Nicotine Patches | Bupropion (Zyban) and Nicotine Patches
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Varenicline (Chantix) | Nicotine Patches | Bupropion (Zyban) and Nicotine Patches
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 0/5 | 0/2 | 0/2

LIMITATIONS AND CAVEATS:
Early termination of the study because of recruitment difficulties lead to insufficient data collection and analysis of primary and secondary outcome measures.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes